CLINICAL TRIAL: NCT01075724
Title: Comparison of a New Patient Warming System Using a Polymer Conductive Warming Under-body and Upper-body Blanket With Forced Air Warming During Surgery
Brief Title: Comparison of a New Patient Warming System Using a Polymer Conductive Warming Under-body and Upper-body Blanket With Forced Air Warming
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Kimberger, Assoc.Prof.PD Dr. MSc, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HDBH3
Record Dates: First submitted 2010-01-25; First posted 2010-02-25 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Hypothermia
Keywords: Perioperative Hypothermia Prevention; Accidental Perioperative Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forced air (Active Comparator): Forced Air Warming
  Interventions: Device: Patient Warming with Forced Air
- Resistive HotDog Warming (Experimental): Warming by resistive Warming
  Interventions: Device: Resistive Warming

INTERVENTIONS:
Device: Patient Warming with Forced Air — Forced Air warming via BairHugger
  Arms: Forced air
Device: Resistive Warming — Resistive Warming via HotDog device
  Arms: Resistive HotDog Warming

SUMMARY:
Intraoperative active warming is usually performed by skin warming. There are several forced-air systems on the market; forced air warming is generally described as the most effective yet feasible method of patient warming.

Augustine Biomedical (Eden Prairie, MN, USA) recently introduced a new patient warming system named "Hot Dog" with an active polymer warming upper-body blanket and a new under-body warming mattress. The polymer-heating devices consist of an electronic regulator and the polymer blankets, which are covered with a washable fabric. Conventional mains power the system. The manufacturer claims, that the new system "Hot Dog" (with combination of under body and upper body warming) is as effective as forced air warming, while not having any disadvantages of the forced air system, like: airborne infection, noise, high power consumption and hard-to-clean hose.

The investigators will compare the new Hot Dog patient warming device combination (under body + upper body) with the established warming system, which blows warm air via a mattress over the body of the patients).

ELIGIBILITY:
Inclusion Criteria:

* The investigators will study 40 patients (18-90 years) undergoing elective orthopedic lower limb surgery at the trauma surgery unit. The patients must have normal weight (20-30 BMI), the duration of surgery should last between 2 - 3 hours.

Exclusion Criteria:

* There will be no other exclusion criteria (except severe peripheral arterial disease in the warmed extremity), as forced air patient warming is routinely used for all patients during this procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Core Temperature at the end of surgery (at time of skin suture) | Single Measurement at Beginning of Skin Suture

SECONDARY OUTCOMES:
Core temperature increase (°C/time) | From Beginning until End of Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Oliver Kimberger, Vienna, Vienna, Austria